CLINICAL TRIAL: NCT06059092
Title: Effects of Three Prophylactic Interventions on French Middle-schoolers' Mental Health: Protocol for a Randomized Controlled Trial
Brief Title: Evaluation of Three School-based Mental Health Preventive Interventions in France
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Nimes (Other)
Responsible Party: Principal Investigator, elodie charbonnier, Lecturer, Qualified to Direct Research, Internal Research Unit Director, University of Nimes
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PrevAdo
Record Dates: First submitted 2023-09-17; First posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Emotional Distress; Functional Impairment; Psychosocial Problem; Wellbeing; User Experience
Keywords: Anxiety; Depression; Psychosocial adjustment; Emotional wellbeing; Social wellbeing; Psychological wellbeing
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: A pre-test assessment will precede all interventions (experimental conditions) and control group sessions delivered simultaneously, and followed by a post-test assessment and and follow-up assessment three months after that.
Masking Description: Participants and their parents will not be aware of precise hypotheses. Nevertheless, for ethical reasons, they are informed that the interventions are meant to improve well-being (before random allocation to control or experimental conditions).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Adapt Module (Experimental): Module targeting reactive adaptation processes
  Interventions: Behavioral: Adapt Module
- Engage Module (Experimental): Module targeting proactive adaptation processes
  Interventions: Behavioral: Engage Module
- Interact Module (Experimental): Module targeting interpersonal adaptation processes
  Interventions: Behavioral: Interact Module
- Control group (Placebo Comparator): Sessions targeting cognitive functions
  Interventions: Behavioral: Control Group

INTERVENTIONS:
Behavioral: Adapt Module — In each intervention, participants will be trained selected psychological skills using cognitive-behavioral-inspired techniques related to coping strategies, locus of control, coping metacognition, positive psychology strategies. Activities will involve brainstorming and exercises based on fictional situations, allowing active participation and reflection as well as feedback from animators and peers. Activities and aids have been designed to meet adolescents' developmental level, concerns and capacities and to support effective learning. Participants will be asked to carry out home tasks to practice learned skills. They will also be provided additional resources related to their module's thematic, accessible through a workbook and a website.
  Arms: Adapt Module
Behavioral: Engage Module — In each intervention, participants will be trained selected psychological skills using cognitive-behavioral-inspired techniques related to goal setting, planning, strengths identification, motivation; goal pursuit metacognition. Activities will involve brainstorming and exercises based on fictional situations, allowing active participation and reflection as well as feedback from animators and peers. Activities and aids have been designed to meet adolescents' developmental level, concerns and capacities and to support effective learning. Participants will be asked to carry out home tasks to practice learned skills. They will also be provided additional resources related to their module's thematic, accessible through a workbook and a website.
  Arms: Engage Module
Behavioral: Interact Module — In each intervention, participants will be trained selected psychological skills using cognitive-behavioral-inspired techniques related to social cognition, assertive communication and conflict resolution, proactive prosocial behaviors, interactional metacognition. Activities will involve brainstorming and exercises based on fictional situations, allowing active participation and reflection as well as feedback from animators and peers. Activities and aids have been designed to meet adolescents' developmental level, concerns and capacities and to support effective learning. Participants will be asked to carry out home tasks to practice learned skills. They will also be provided additional resources related to their module's thematic, accessible through a workbook and a website.
  Arms: Interact Module
Behavioral: Control Group — Sessions will be devoted to serious game training cognitive and executive functions through individual and group activities based on board games.
  Arms: Control group

SUMMARY:
To meet adolescents' needs regarding mental health vulnerability, this study aims to propose and evaluate three original school-based preventive interventions delivered to French 13y-adolescents, with respect to their effects on mental health outcomes, as well as users' experiences of intervention, evaluated through questionnaires. Based on cognitive-behavioral therapies (CBT) techniques, these interventions target three strategic process areas: reactive adaptation, proactive adaptation, and interpersonal adaptation. Their effectiveness will be evaluated through a four-arm randomized controlled trial, conducted in an ecological context. Intra-group and inter-group comparisons will be carried out for our different variables of interest, namely targeted psychological processes, levels of distress, functional impairment, and well-being, and user experience indicators of acceptability, utility, and usability.

DETAILED DESCRIPTION:
The three interventions will be delivered in school facilities, during school time, with 4th-grade middle school students, by one psychologist trained in CBT and one undergraduate student in clinical psychology in CBT. They involve participating in three one-hour weekly sessions, plus one booster sessions one month later. These three programs have been designed based on pre-existing knowledge about adolescents and their cognitive-motivational mechanisms, in order to promote their learning and receptiveness to interventions, and include group and individual activities meant to improve key psychological processes. The control group will consist of the same number of sessions of identical length as experimental conditions, dedicated to serious games meant to work on cognitive functions (attention, memory, logical reasoning).

For all participants, several indicators of mental health and of cognitive-behavioral processes will be measured through validated self- and parent-reported questionnaires, and completed by user experience questionnaires. Mixt linear models or non-parametric equivalent tests will be conducted to test hypotheses (i.e., positive change in all outcomes following interventions in the experimental conditions, not observed in the participants of the control group).

The interventions are preventive and will not target adolescents at risk for psychopathological conditions. Nevertheless, it is possible that at-risk individuals are enrolled in the sample. To meet special needs of some participants, from the beginning of the study, professional mental health resources (phone number, websites, institutions) will be provided to all participants. A clinical psychologist (one of tthe animator) will be available for students who would ask for individual appointments by handling duty periods in school facilities two hours a week during the interventions.

ELIGIBILITY:
Inclusion Criteria:

* being enrolled in one of the middle school involved in the study
* parent and student consent for participation
* parent and student proficiency in French

Exclusion Criteria:

* absence or withdrawal of consent (parent or student)
* missing more than 1 in 4 sessions

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2023-11-06 (Estimated); Primary Completion 2023-12-22 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
General distress | Post-test 3 weeks after pre-test, follow-up 3 months after post-test
  Anxiety and depressive symptoms (Hospital Anxiety and Depression Scale). A high score on each subscale (anxiety symptoms subscale, 7 items, and depression symptoms subscale, 7 items), ranging from 0 to 21, indicates a high level of anxiety or depression. A high composite score (addition of scores yielded by the 2 subscales), ranging from 0 to 42, indicates a high level of general distress.
Wellbeing | Post-test 3 weeks after pre-test, follow-up 3 months after post-test
  Psychological, social and emotional well-being (Mental Health Continuum-Short Form). A high score on each emotional, social, and psychological wellbeing subscales, ranging from 3 or 6 to 18 or 36 depending on subscales, indicate a high level of each kind of wellbeing. A high composite score (ranging from 14 to 84) indicates a high level of general wellbeing.
Functional impairment | Post-test 3 weeks after pre-test, follow-up 3 months after post-test
  Functional impairment in school, social, personal, domestic areas (Work and Social Adjustment Scale for Youth; WSAS-Y). A high score (ranging from 0 to 40) indicates a high level of functional impairment across these life areas.
Psychosocial difficulties | Post-test 3 weeks after pre-test, follow-up 3 months after post-test
  Psychosocial difficulties of various internalized and externalized natures, measured by the Pediatric Symptom Checklist (PSC). A high score (ranging from 0 to 70) indicates a high level of psychosocial difficulties.
Type of coping strategies | Post-test 3 weeks after pre-test, follow-up 3 months after post-test
  Brief-COPE. A high score on each of the 14 strategies subscales (e.g., denial, acceptance, planning, disengagement), ranging from 2 to 8, indicates a frequent use of each strategy.
Coping Flexibility | Post-test 3 weeks after pre-test, follow-up 3 months after post-test
  Coping Flexibility Scale. A high score (ranging from 7 to 28) indicates a high level of coping flexibility.
Tendency to engage in committed action | Post-test 3 weeks after pre-test, follow-up 3 months after post-test
  Willingness and Action Measurement for Children and Adolescents (WAM-C/a), Action subscales. A high score (ranging from 9 to 45) indicate a high tendency do carry out actions related to important personal values despite negative feelings.
General Self-Efficacy | Post-test 3 weeks after pre-test, follow-up 3 months after post-test
  General Self Efficacy scale-Short-form (S-GSES). A high score (ranging from 3 to 15) indicates a high level of general self-efficacy.
Assertiveness in interaction | Post-test 3 weeks after pre-test, follow-up 3 months after post-test
  Ability to express feelings and opinions to others and to respect others (Assertiveness Formative Questionnaire)

SECONDARY OUTCOMES:
User experience questionnaire | Post-test 3 weeks after pre-test, follow-up 3 months after post-test
  Participants' perceived utility, acceptability, usability and general appreciation of the interventions
Sociodemographic data 1 | Post-test 3 weeks after pre-test, follow-up 3 months after post-test
  Adolescents' gender (qualitative questionnaire, unscored)
Sociodemographic data 2 | Post-test 3 weeks after pre-test, follow-up 3 months after post-test
  Adolescents' age (questionnaire, unscored)
Sociodemographic data 3 | Post-test 3 weeks after pre-test, follow-up 3 months after post-test
  Adolescents' current and previous diagnoses and treatments qualitative (qualitative questionnaire, unscored)
Sociodemographic data 4 | Post-test 3 weeks after pre-test, follow-up 3 months after post-test
  Family status (qualitative questionnaire, unscored)
Sociodemographic data 5 | Post-test 3 weeks after pre-test, follow-up 3 months after post-test
  Home income (questionnaire, unscored)
Sociodemographic data 6 | Post-test 3 weeks after pre-test, follow-up 3 months after post-test
  Parents' gender, profession, education level (qualitative questionnaire, unscored)

CONTACTS AND LOCATIONS:
Overall Officials: Elodie Charbonnier, MCF HDR, Principal Investigator — UPR APSY-v University of Nîmes
Locations (2):
- France (2):
  - Institut Valsainte, Nîmes, Gard
  - Collège Révolution, Nîmes, Gard

IPD SHARING:
Plan to Share IPD: Undecided